CLINICAL TRIAL: NCT02707003
Title: A Multi-Center Pilot Observational Trial to Quantify the Potential Clinical Utility of Capnography in the PACU
Brief Title: Clinical Utility of Capnography in the PACU( Post-anaesthesia Care Unit)
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVMOPO0526
Record Dates: First submitted 2016-03-07; First posted 2016-03-11 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Respiratory Depression
Keywords: Post-operative respiratory distress
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: Yes

GROUPS / COHORTS (2):
- AZ PACU: Observation of standard of care with capnography blinded
- TWH PACU: Observation of standard of care with capnography blinded

SUMMARY:
Multi-center observational trial with study device blinded in order to assess in parallel standard monitoring and intervention practices related to management of respiratory compromise in the post-anaesthesia care unit (PACU)

DETAILED DESCRIPTION:
All Study device information is blinded to medical staff but the Study Coordinator will have full access to device measurements, alarms, notification and events via a local Wi-Fi hub sent to a portable tablet. The tablet Case Report Form (CRF) will allow all observation be inserted with a time stamp on the electronic device data. In addition, all electronic data will be collected from the bedside monitor.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥ 18 years of age
2. ASA Score II - IV (American Society of Anaesthesiologists Score)
3. Patients booked for a surgical procedure requiring general anesthesia care
4. Expected duration of general anesthesia to be > 1.5 hours
5. Expected to receive intraoperative opioids
6. Expected to be transferred to the PACU from the operating room
7. Patients with an expected duration in the PACU ≥ 45 minutes
8. Expected to be transferred from the PACU to an in-patient setting

Exclusion Criteria:

1. Patients expected to be discharged from the hospital when discharged from the PACU
2. Subjects who will have oral/nasal surgery that may prevent wearing an oral/nasal capnography sampling filterline.
3. Subjects with a history of severe contact allergies that may cause a reaction to standard adhesive materials found in pulse oximetry sensors.
4. Patients with skin lesions or physical deformities that would prevent the application of finger sensors for optimal performance.
5. A female known to be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults booked for a surgical procedure that meet the I/E criteria and willing to provide consent for observation in the PACU and chart review 24 hours post PACU discharge.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2016-02; Primary Completion 2017-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Frequency of Respiratory Adverse Events in the PACU identified by capnography | Up to 2 hours in the PACU
  Identification by blinded capnography to understand the ventilation challenges of patient in the PACU during standard of care that does not include capnography. First tier is RN (Registered Nurse) level of notification for early intervention and second tier is level at which covering MD (Medical Doctor) might request notification:
  1. High Respiration Rate >25 bpm for > 15 seconds (tier one) and >30 bpm for more than 30 seconds (tier two)
  2. Low Respiration Rate < 8 bpm for more than 15 seconds and < 6 bpm for more than 30 seconds
  3. High end tidal CO2 (EtCO2) > 55 mmHg for > 15 seconds and > 60 mmHg for more than 30 seconds
  4. Low EtCO2 < 25 mmHg for > 15 seconds and < 25 mmHg for more than 30 seconds
  5. High Heart Rate > 120/min for 15 seconds and >120/min for 30 seconds
  6. Low Heart Rate < 40/min for 15 seconds and < 40/min for 30 seconds
  7. SpO2 (oxygen saturation by pulse oximetry) /Hypoxemia < 90% for more than 15 seconds and< 90% for more than 30 seconds

SECONDARY OUTCOMES:
Frequency of Critical Adverse Events (CRAE) | PACU and 24 hours post PACU
  Critical CRAE in the PACU or in 24 hour post PACU chart review:
  1. Narcotic overdose that required an Opioid reversal
  2. Partial airway obstruction that required an NMBA (neuromuscular blocking agent) antagonist
  3. Respiratory Insufficiency that would require Non-invasive positive pressure ventilation, ambu bag mask assisted ventilation
  4. Respiratory failure that would Invasive mechanical ventilation
  5. Upper airway obstruction requiring airway support measures (oral or nasal) such as intubation, LMA (laryngeal mask airway), or airway
  6. Respiratory insufficiency/failure that would require a transfer to the ICU
  7. Cardiopulmonary arrest
  8. Death due to respiratory/pulmonary related complications Other (free text that might capture aspiration, pneumothorax)
Ventilation insufficiency on transfer from the PACU | At PACU discharge
  Population of patients leaving the PACU in early stage ventilation respiratory insufficiency as defined as etCO2 ≤ 25 mmHg or etCO2 ≥55 mmHg combined with low RR (respiratory rate) and hypotension within 15 minutes before transport out of the PACU.

CONTACTS AND LOCATIONS:
Overall Officials: Peter R Lichtenthal, MD, Principal Investigator — Banner University Medical Center; Francis F Chung, MBBS FRCPC, Principal Investigator — University Health Network, Toronto
Locations (2):
- Banner University Medical Center, Tucson, Arizona, United States
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kanaparthi A, Chung F, Lichtenthal PR, Sprung J, Weingarten TN. PRODIGY score predicts respiratory depression in the post-anesthesia care unit: A post-hoc analysis. Biomol Biomed. 2024 Oct 17;24(6):1662-1668. doi: 10.17305/bb.2024.10585. PMID 38843498
- [Derived] Chung F, Wong J, Mestek ML, Niebel KH, Lichtenthal P. Characterization of respiratory compromise and the potential clinical utility of capnography in the post-anesthesia care unit: a blinded observational trial. J Clin Monit Comput. 2020 Jun;34(3):541-551. doi: 10.1007/s10877-019-00333-9. Epub 2019 Jun 7. PMID 31175500
- See also: Post Study Publication — https://pubmed.ncbi.nlm.nih.gov/31175500/